## NAME OF THE STUDY:

Evaluation of the effectiveness of psychoeducational training given to nurses working in a psychiatric clinic: Randomized controlled study.

## STUDY PROTOCOL

The research is a randomized controlled experimental study. The sample of the study consisted of a total of 78 nurses working in the psychiatry clinic of Etlik City Hospital, 39 of which were in the experimental group and 39 in the control. "Psychoeducational knowledge and skills development training of nurses working in psychiatric clinic" was given to the experimental group as a total of 4 sessions, each session being two sessions of 50 minutes. The data of the study were collected with the "Personal Information form", "The form for evaluating the knowledge level of the nurses working in the psychiatry clinic about psychoeducation" and "The scale of perception of competence in developing and implementing a psychoeducational program".

## STATISTICAL ANALYSIS PLAN

Percentage, arithmetic mean, T test in independent samples, One Way ANOVA, Wilcoxon test, Bonferroni test were used in SPSS 26.0 statistical program for data analysis. p<0.05 statistical significance condition was sought.

## INFORMED CONSENT FORM

A research has been planned in order to increase the competence perceptions of nurses working in psychiatric clinics for psychoeducation planning and implementation.

The aim of the study is to improve the competence perceptions of psychoeducational planning and implementation of nurses working in psychiatric clinics. We invite you to participate in this research to be conducted. If you agree to participate in the study, you will not be charged any fee and you will not be paid any fee for participating. Your information will be kept confidential, but it can be examined by the ethics committee or official authorities if necessary. Participation in the study depends entirely on your volunteering. You also have the right to withdraw your consent at any stage of the study without being subject to any penalties or sanctions. First of all, we want to inform you about the study, if you want to participate in the research after reading and understanding this information, please sign the form. If you agree to participate in the study, you will be asked to fill out the questionnaire form created by our researchers. Then, the training program consisting of a total of four sessions, one per week, will be given in the form of 2 sessions of 50 minutes. Subject headings, date time will be given to you in writing. After all the trainings are completed, the forms filled in at the beginning of the training will be filled out again. For questions about the study, you can call Nermin Erdogan's phone number 0533 468 79 22. Thank you for your contributions in advance.

PHD Nurse Nermin Erdogan

| The Participant |
|-----------------|
| name surname: |
| History: |
| Signature: |

PARTICIPANT STATEMENT

I was invited by Mr. Nermin Erdogan as a "participant" by transferring the above information

about the research to be conducted in order to evaluate the "evaluation of psychoeducational

planning and implementation competency perceptions of nurses working in a psychiatric

clinic to improve their education".

I am not under any financial responsibility for the research. No payment will be paid to my

side. During the conduct of the research, I may leave the research without giving any reason. I

have been informed that my personal information will be protected when the research results

are used for scientific purposes. I know that if I have any problems related to the

implementation of the research, I can call the responsible researcher Nermin Erdogan from

the phone number forwarded to me. Before starting the research, I read the written

information and listened to the oral explanations. I agree to participate in this research with

my consent, without any pressure or coercion and voluntarily.

The Participant's Name-Surname:

Address:

The Wire:

Date and Signature:

Name-Surname of the researcher who made the statements: Nermin Erdogan

Address: Etlik City Hospital Psychiatric Clinic

Tel: 0334687922

Date and Signature: